CLINICAL TRIAL: NCT00031473
Title: A Randomized Phase III Study to Evaluate the Safety and Efficacy of Ribavirin Inhaled Solution in Preventing Progression of Upper Respiratory Tract Respiratory Syncytial Virus Infection to RSV Pneumonia in Blood and Bone Marrow Transplant (BMT) Recipient
Brief Title: Ribavirin to Prevent RSV Pneumonia in Bone Marrow Transplant Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 97-038; NCT00001098 (obsolete NCT alias)
Record Dates: First submitted 2002-03-06; First posted 2002-03-07 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2003-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Ribavirin; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Ribavirin

INTERVENTIONS:
Drug: Virazole (Ribavirin) Inhalation Solution

SUMMARY:
The purpose of this study is to test the safety and effectiveness of ribavirin, administered as an aerosol, in preventing progression of upper respiratory tract RSV infection to RSV pneumonia in bone marrow and peripheral blood transplant recipients.

DETAILED DESCRIPTION:
The study enrolls 90 transplant recipients with positive nasal/throat culture specimens for Respiratory Syncytial Virus (RSV) infection. Patients are randomized into one of two groups: investigational treatment or standard treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* 2 years of age or older.
* Are not pregnant or breast-feeding and agree to use a reliable birth control method for the duration of the study.
* Are a blood or bone marrow transplant recipient.
* Have evidence of upper respiratory tract infection.
* Have nasopharyngeal-throat samples positive for RSV.

EXCLUSION CRITERIA:

* Are known to be HIV positive.
* Have pneumonia.
* Require a ventilator to breathe.
* Are pregnant.
* Are breast-feeding and are unwilling to stop breast-feeding.
* Are receiving treatment with certain other drugs for RSV.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90
Dates: Start 1997-11; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama at Birmingham (CASG), Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - J. Whitcomb Riley Hosp for Chldrn - Indianapolis, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - St. Luke's Hospital (Kansas City, MO), Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - SUNY Upstate Medical University, Syracuse, New York